CLINICAL TRIAL: NCT05313204
Title: Physiological Responses to Exercise During Pregnancy in People With Multiple Sclerosis
Brief Title: Exercise and Pregnancy in People With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00095678
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis; Pregnancy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant with Multiple Sclerosis: Pregnant individuals (> 13 weeks) with a Multiple Sclerosis diagnosis.
  Interventions: Other: Moderate-intensity cardiovascular exercise
- Pregnant without Multiple Sclerosis: Pregnant individuals (> 13 weeks) without Multiple Sclerosis.
  Interventions: Other: Moderate-intensity cardiovascular exercise
- Postpartum with Multiple Sclerosis: Postpartum individuals (< 1 year since delivery) with a Multiple Sclerosis diagnosis.
  Interventions: Other: Moderate-intensity cardiovascular exercise
- Postpartum without Multiple Sclerosis: Postpartum individuals (< 1 year since delivery) without Multiple Sclerosis.
  Interventions: Other: Moderate-intensity cardiovascular exercise

INTERVENTIONS:
Other: Moderate-intensity cardiovascular exercise — The participant will be instructed to first rest quietly for 10 minutes wearing a heart rate monitor. The participant will then be instructed to exercise at an intensity of 60-70% heart rate reserve (HRR) for 20 minutes. The participant may choose any kind of cardiovascular exercise modality they prefer, as long as the exercise will meet the prescribed intensity. Following exercise, participants will rest quietly for 10 minutes wearing the heart rate monitor.

SUMMARY:
The purpose of this study is to examine acute physiological responses to exercise and activity patterns of people with multiple sclerosis (MS) during pregnancy and postpartum.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an inflammatory autoimmune condition of the central nervous system, which causes demyelination of axons, and largely affects females aged 20-40 years. However, knowledge gaps surrounding MS in pregnancy and postpartum remain. Particularly, no research has examined the effects of exercise or physical activity patterns, in people with MS throughout pregnancy and postpartum. Current guidelines for exercise in pregnancy note that people with impairments may safely meet activity recommendations; however, medical consultation is recommended. This study aims to provide information regarding the physiological responses to exercise, as well as the physical activity patterns of pregnant and postpartum people with MS.

Numerous studies have found pregnant individuals with MS experience reduced rates of relapse (periods of symptom exacerbation) during pregnancy, most significantly in the third trimester. Additionally, increased rates of relapse in the three months following delivery among people with MS has been commonly observed. These unique periods combined with maternal adaptations during and following pregnancy may impact responses to exercise during and following pregnant in people with MS. To our knowledge, no research has investigated the physiological responses to exercise nor physical activity patterns in individuals with MS during or following pregnancy. These data will be used to develop prospective interventions aimed at determining the causal links between adaptations to pregnancy and postpartum and exercise tolerance in people with MS. They will also be a critical first step towards the eventual development of evidence-based guidelines for pregnant and postpartum people with MS.

Pregnant and postpartum individuals will be sent the equipment and questionnaires needed to participate in this virtual study. Participants will complete a 20-minute moderate-intensity exercise bout (60-70% heart rate reserve) using their own cardiovascular exercise equipment or walking outside. During exercise, participants will wear a heart rate monitor to measure heart rate prior to, during and following exercise, as well as complete a fatigue assessment prior-to, immediately, and 30- and 60-minutes following exercise. Additionally, participants will wear a continuous glucose monitor (Freestyle Libre Pro) throughout the exercise and for seven days following exercise. Participants will also wear two non-invasive activity monitoring devices that measure their activity and sedentary time for seven full days. Lastly, participants with MS will track their MS symptoms for seven full days. These data will have implications in understanding the acute cardiovascular response to moderate-intensity exercise among pregnant and postpartum people with MS. This is an important first step in understanding the benefits of pre- and postnatal physical activity among people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis diagnosis
* Pregnant with a single baby (> 13 weeks) or Postpartum (< 1 year since delivery)
* Free of cardiovascular disease

Exclusion Criteria:

* Pregnant individuals who have absolute contraindications to exercise as outlined by the Canadian Guidelines for Exercise in Pregnancy PARMed-X questionnaire OR relative contraindications that prevent them from exercise as confirmed by their medical professional.
* High-order pregnancies, e.g. twins or above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant (> 13 weeks) and postpartum (< 1 year since delivery) individuals with Multiple Sclerosis.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | 40 minutes
  Resting heart rate will be measured immediately prior-to exercise. Change in heart rate will be measured during and following exercise.
Fatigue | 10 minutes
  Fatigue will be assessed immediately before, immediately following, 30- and 60-minutes following exercise using the Visual Analog Scale to Assess Fatigue Severity.
Physical activity and sedentary behaviour | 7 days
  Participants will wear an accelerometer and activPAL (Actigraph wGT3X-BT Monitor, Actigraph LLC; activPAL, PAL Technologies Ltd.) for seven consecutive days and nights to record 24-hour physical activity and sleep/wake measurements.

SECONDARY OUTCOMES:
Glucose | 40 minutes
  Glucose response to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Margie Davenport, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada